CLINICAL TRIAL: NCT05349877
Title: Efficacy of a Brief, Self-guided, On-line, Writing Intervention to Improve Mental Health Outcomes Among Sexual and Gender Minorities: a Randomized Controlled Trial.
Brief Title: Efficacy of a Brief Intervention to Improve Sexual and Gender Minorities' Mental Health: Randomized Controlled Trial.
Acronym: ESCREVA-SE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PUCRSBR-10098; 39059120.0.0000.5336 (Other: Brazil's Plataforma Brasil CAAE)
Record Dates: First submitted 2022-03-11; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2021-10

CONDITIONS: Depression; Anxiety; Psychological Distress; Social Phobia; Post Traumatic Stress Disorder; Suicidal Ideation; Sex, Unsafe; Discrimination, Social; Behavior, Risk; Self Esteem
MeSH Terms: conditions — Depression; Anxiety Disorders; Phobia, Social; Stress Disorders, Post-Traumatic; Suicidal Ideation; Unsafe Sex; Social Discrimination; Risk-Taking

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, clinical trial assessing the efficacy of a brief, unsupervised, self-guided psychological intervention targeting sexual and gender minorities' mental health.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Expressive writing (Experimental): Participants will be invited to join three writing activities, lasting 20 minutes daily in D1, D3, and D5 of the same week. For example, to write about a difficult or painful experience related discrimination and their feelings about it.
  Interventions: Behavioral: Expressive writing
- Self-affirmation (Experimental): Aiming to build self-efficacy, participants will be invite to writing, during 20 minutes daily in D1, D3, and D5 of the same week, a letter to a sexual and gender minority peer suffering from stigma and discrimination.
  Interventions: Behavioral: Self-affirmation
- Placebo (Placebo Comparator): Participants will be instruct to write about their daily routine, during 20 minutes daily in D1, D3, and D5 of the same week.
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Expressive writing — Write, continuously for 20 minutes, about deepest emotions and thoughts concerning experiences of minority stress, exploring a particular event and how it has affected the participant.
  Arms: Expressive writing
Behavioral: Self-affirmation — Write, continuously for 20 minutes, about values the participant think is important to overcome experiences of minority stress.
  Arms: Self-affirmation
Behavioral: Placebo — Write, continuously for 20 minutes, about their daily routine, without expressing feelings and deep thoughts about it.
  Arms: Placebo

SUMMARY:
Experiences of violence, from micro to physical aggressions, have a deleterious impact on mental health. According to the Minority Stress Theory, unfavorable social conditions (such as anticipated and experienced discrimination and internalized homophobia), mediated by resilience strategies, can lead to mental health or illness. Sexual and gender minorities (SGM) face stigma and discrimination aggravating multiple aspects of their lives: from school drop-out to halting health care access. SGM reveal avoiding medical assistance for fear of discrimination while health professionals disclose feeling unprepared to handle SGM health needs. There are two main challenges: 1) developing specific psychological interventions to reduce the impact of stigma and discrimination on SGM' mental health; and 2) training public health professionals to properly address SGM needs. Therefore, the present trial aims to assess the efficacy of a brief, self-guided, on-line, asynchronous and unsupervised psychological intervention in improving SGM' mental health.

ELIGIBILITY:
Inclusion Criteria:

* Self-identity as sexual and gender minority.
* Being older than 16 years old.
* Have a stable on-line connection for, at least, 20 minutes in a place where won't be disturbed.
* Reports, in the baseline survey, previous experiences of discrimination, having depression or anxiety symptoms.
* Currently living in Rio Grande do Sul.

Exclusion Criteria:

* Disagrees with the consent form.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2022-06-10 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline depression at 3 and 6 moths after the intervention. | Baseline (T0), one week after the intervention (T1), three months after the intervention (T2), and six the intervention (T3).
  Assessed using the Center for Epidemiologic Studies - Depression (CES-D). CES-D is composed of 20 items. The final score ranges from 0 to 60 points. Originally, the cutoff point of the CES-D scale to identify the presence of depressive symptoms is equal or higher 16 points. However, when considering Brazilian samples, the cutoff point of equal or higher 12 points was proposed.
Change from baseline anxiety at 1 week, and 3 and 6 moths after the intervention. | Baseline (T0), one week after the intervention (T1), three months after the intervention (T2), and six the intervention (T3).
  Evaluated using the Generalized Anxiety Disorder 7-item (GAD-7). The GAD-7 consists of 7 questions based in part on the DSM-IV criteria for GAD and reflects the frequency of symptoms during the preceding 2-week period. The GAD-7 requires approximately 1-2 minutes to administer and for each symptom queried provides the following response options: "not at all," "several days," "over half the days" and "nearly every day" and these are scored, respectively, as 0, 1, 2 or 3. A score of 10 or greater on the GAD-7 represents a reasonable cut point for identifying cases of GAD.
Change from baseline social phobia at 1 week, and 3 and 6 moths after the intervention. | Baseline (T0), one week after the intervention (T1), three months after the intervention (T2), and six the intervention (T3).
  Evaluated using the Social Avoidance and Distress Scale (SADS). SADS is a 28 item true/false scale that measures measures aspects of social anxiety including distress, discomfort, fear and avoidance. A total score on the SADS is obtained based on the answers to the true/false questions. Higher scores indicate greater social anxiety.
Change from baseline post-traumatic stress at 1 week, and 3 and 6 moths after the intervention. | Baseline (T0), one week after the intervention (T1), three months after the intervention (T2), and six the intervention (T3).
  Post-Traumatic Stress Disorder Checklist - Civilian Version (PCL-C). The PCL-C is a 17-item self-report checklist of PTSD symptoms based closely on the DSM-IV criteria. The score consists in adding up all items from each of the 17 items for a total severity score (range = 17-85). The cut off 17-29 shows little to no severity, 28-29 suggests some PTSD symptom, 30-44 moderate to moderately high severity of PTSD symptoms, and 45-85 high severity of PTSD symptoms.
Change from baseline on suicide ideation at 3 and 6 moths after the intervention. | Baseline (T0), three months after the intervention (T2), and six the intervention (T3).
  Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a clinically-validated screening tool that healthcare providers use to screen for depression, and also to diagnose and monitor the severity of the condition. A PHQ-9 score total of 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression.
Change from baseline on substance use at 3 and 6 moths after the intervention. | Baseline (T0), three months after the intervention (T2), and six the intervention (T3).
  Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) is an 8 questions tool that detects substance use and related problems. A 'global continuum of risk score' (or total substance involvement) is calculated by the addition of all items for all substances on the ASSIST and has a maximum score of 208.
Change from baseline on sex risk behaviors at 3 and 6 moths after the intervention. | Baseline (T0), three months after the intervention (T2), and six the intervention (T3).
  Inquired using yes-no questions concerning unprotected intercourse and multiple sex partners, as well as the Perceived Risk of HIV Scale. Perceived Risk of HIV Scale is a self-report 8-item measure developed to assess how people think and feel about their risk of HIV infection based on their previous sexual behavior and covering several dimensions of perceived HIV risk. Higher scores are associated with a greater number of sex partners, episodes of unprotected sex and having sex while high.

SECONDARY OUTCOMES:
Change from baseline on resilience at 1 week, and 3 and 6 moths after the intervention. | Baseline (T0), one week after the intervention (T1), three months after the intervention (T2), and six the intervention (T3).
  Wagnild and Youngs's Resilience Scale that has presented the following scoring for the total score: 25-100 = Very low, 101-115 = Low, 116-130 = On the low end, 131-145 = Moderate, 146-160 = Moderately high, and 161-175 = High.
Change from baseline on self-esteem at 1 week, and 3 and 6 moths after the intervention. | Baseline (T0), one week after the intervention (T1), three months after the intervention (T2), and six the intervention (T3).
  Rosenberg Self-Esteem Scale. The scale ranges from 0-30. Scores between 15 and 25 are within normal range; scores below 15 suggest low self-esteem.

IPD SHARING:
Plan to Share IPD: No